CLINICAL TRIAL: NCT01018329
Title: Multimodality Statistical Model of Early Response of High Grade Glioma to Radiation Therapy
Brief Title: Magnetic Resonance Imaging in Evaluating Response to RadiationTherapy in Patients With High Grade Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 12309
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Brain Tumor
Keywords: Adult Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Patients undergo multimodality MRI imaging at baseline, weeks 1, 2, 3, 5, and 6 and then 4-6 weeks after completion of radiation therapy.Patients undergo MRI imaging at baseline, weeks 1, 2, 3, 5, 6 and then 6 weeks after radiation therapy.
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Diffusion Tensor Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging; Procedure: Dynamic Contract-Enhanced magnetic resonance imaging; Procedure: Diffusion-weighted magnetic resonance imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging
  Other Names: MRI,NMR imaging, NMRI, nuclear magnetic resonance imaging
Procedure: Diffusion Tensor Imaging
Procedure: Magnetic Resonance Spectroscopic Imaging
  Other Names: 1H-nuclear magnetic resonance spectroscopic imaging, Proton Magnetic Resonance Spectroscopic Imaging
Procedure: Dynamic Contract-Enhanced magnetic resonance imaging
  Other Names: DCE-MRI
Procedure: Diffusion-weighted magnetic resonance imaging
  Other Names: diffusion-weighted MRI

SUMMARY:
RATIONALE: Diagnostic procedures, such as magnetic resonance imaging, may help doctors predict a patient's response to treatment and help plan the best treatment. PURPOSE: This clinical trial is studying magnetic resonance imaging in response to radiation therapy in patients with high grade glioma.

DETAILED DESCRIPTION:
Detailed DescriptionOBJECTIVES:

I. To develop a multimodality statistical model to act as a surrogate marker scheme of early changes in high grade glioma patients undergoing radiation therapy, using conventional MRI, MR diffusion tensor imaging, perfusion, permeability, and spectroscopic imaging while incorporating the radiation dose calculations delivered locally and the results of a clinical questionnaire into the model.

II. To assess treatment response to tumor and normal tissue changes. OUTLINE: Patients undergo multimodality MRI imaging at baseline, weeks 1, 2, 3, 5, and 6, and then 4-6 weeks after completion of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated for diagnosed with high grade glioma (WHO grade III or IV) at the University of Pennsylvania Medical Center who will be undergoing radiation therapy to the brain
* Patient or legal representative able to provide written informed consent
* Adult males and nonpregnant females

Exclusion Criteria:

* Vulnerable populations as specified (including pregnant patients, prisoners, patients with pacemakers or metallic implants)
* Patients with renal failure
* Patients with any condition considered a contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Early brain tumor response

SECONDARY OUTCOMES:
Early therapeutic-induced changes in normal surrounding brain

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States